CLINICAL TRIAL: NCT04905758
Title: Soft and Hard Tissues Evaluation Around Immediately Placed New Implant Design: Randomised Clinical Study
Brief Title: Soft and Hard Tissues Evaluation Around Immediately Placed New Implant Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, lecturer of oral medicine and periodontology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: assmortada2020
Record Dates: First submitted 2021-05-26; First posted 2021-05-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Peri-implant Mucositis; Dental Implant Failed
Keywords: platform switched implants; platform matched implants
MeSH Terms: interventions — Dental Implant-Abutment Design

STUDY DESIGN:
Intervention Model Description: Maxi-Z plus dental implant
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxi-Z plus dental implant (Experimental): platform switched dental implants
  Interventions: Procedure: platform switching
- Maxi-Z dental implant (Active Comparator): platform matched dental implants
  Interventions: Procedure: platform amtching

INTERVENTIONS:
Procedure: platform switching — reduced implant abutment interface
  Arms: Maxi-Z plus dental implant
Procedure: platform amtching — matched implant abutment interface
  Arms: Maxi-Z dental implant

SUMMARY:
patients were randomly divided into Maxi-Z plus dental implant group versus Maxi-Z implant group

DETAILED DESCRIPTION:
after tooth extraction implants will be placed immediately and provisional restoration will be placed in both groups to detect the advantaged and drawbacks of newly designed Maxi-Z plus dental implant versus Maxi-Z dental implant

ELIGIBILITY:
Inclusion Criteria:

* good health
* unrestorable, periodontal healthy teeth

Exclusion Criteria:

* systemic disease
* periodontal disease
* presence of abscess

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Implant mobility using Periotest M | 12 months
  Periotest M values range from (-8 to 0). high values represent loose implant, while osseointegrated implants showed low values
marginal bone level | 12 months
  measured in mm using X-ray

SECONDARY OUTCOMES:
pink estheic score | 12 months
  from 0-12. 0 means bad aesthetic of soft tissue. 12 means the ultimate aesthetics of soft tissue

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after research results publishing will decide
Supporting Information: Study Protocol
Time Frame: by the end of August 2021 for 6 months
Access Criteria: open access